CLINICAL TRIAL: NCT01979666
Title: the Effect of a Nitrate Patch on the Healing Process of AVN of the Knee
Brief Title: Nitrate Patch Use as Treatment of Knee AVN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit patients
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof.Avi Livneh, head of internal medicine ward F, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-12-9707-AL-CTIL
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Necrosis, Avascular, of Bone
Keywords: Knee AVN, Nitrates
MeSH Terms: conditions — Osteonecrosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): the patients that will get a nitrate patch
  Interventions: Drug: nitrate patch; Device: MRI scan
- control group (Placebo Comparator): the patients that will get the placebo patch
  Interventions: Drug: placebo patch; Device: MRI scan

INTERVENTIONS:
Drug: nitrate patch — patients in the study group will get a nitrate patch
  Arms: study group
Drug: placebo patch — control group patients will get a placebo patch
  Other Names: placebo
  Arms: control group
Device: MRI scan — MRI scan after 6 weeks of treatment
  Other Names: MRI

SUMMARY:
The pathogenesis of AVN includes a defective blood supply to the knee joint. Local nitrates induce peripheral vasodilation and may improve blood supply to the affected tissue.

This study aims to test whether the use of a nicotine patch may accelerate the healing process from AVN of the knee.

DETAILED DESCRIPTION:
The main purpose of this study is to examine whether treatment with a local nitrate patch will improve MRI findings and clinical outcomes in patients with AVN of the knee.

This is a double-blind prospective study that will include 50 adult volunteers, randomly assigned to a "nitrate" group that will be given a nitrate patch, and a "placebo" group that will be given a placebo patch.

The following outcomes will be measured:

* MRI findings before and after the patch treatment
* Use of analgesics
* Subjective pain relief.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18-80 y.o)
* diagnosis of AVN according to MRI

Exclusion Criteria:

* Terminal illness
* Cognitive impairment / any condition disturbing informed concent.
* Nitrate intolerance
* Patients using Cyclic GMP inhibitiors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Reduction in bone substrate edema | 6 weeks
  the area and percent of the knee which the edema involves

SECONDARY OUTCOMES:
other MRI changes | 6 weeks
  reduction of subchondral fracture resolution of accompanied findings presence of femoral head or condyle flattening
analgesics use | 6 weeks
  according to the patient's self report
pain severity | 6 weeks
  according to a visual analouge scale

CONTACTS AND LOCATIONS:
Overall Officials: avi livneh, Principal Investigator — Sheba Medical Center; arik asman, MD, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel